CLINICAL TRIAL: NCT00234338
Title: Prospective Post-Marketing Surveillance Study of Prevenar in High-Risk Children Aged 2 to 5 Years
Brief Title: Study Evaluating Prevenar in High-Risk Children
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 101850
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Pneumococcal Disease
Keywords: Children; Vaccine; Prevenar
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to estimate the local and systemic tolerability of Prevenar in children ages 2 to 5 years old in usual care settings.

ELIGIBILITY:
Inclusion Criteria:

* High-risk children ages 2 to 5 years old

Exclusion criteria:

* Prior administration of Prevenar
* Prior and/or concurrent administration of 23 vPs vaccine

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2005-10; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com
Locations (1):
- Frankfurt, Germany